CLINICAL TRIAL: NCT05033795
Title: Metabolomic Evaluation of the Impact of Rocchetta Water on the Skin of Healthy Patients Through the Innovative Method of Artificial Intelligence.
Brief Title: Metabolomic Evaluation of the Impact of Acqua Rocchetta on the Skin of Healthy Patients.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: I.R.C.C.S Ospedale Galeazzi-Sant'Ambrogio (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Health Services Research
Other Study IDs: VALORE
Record Dates: First submitted 2021-06-14; First posted 2021-09-05 (Actual); Last update posted 2021-09-05 (Actual); Status verified 2021-08

CONDITIONS: Skin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Water A (Experimental): 2 L of water A per day
  Interventions: Dietary Supplement: Water A
- Water B (Other): 2 L of water B per day
  Interventions: Dietary Supplement: Water B

INTERVENTIONS:
Dietary Supplement: Water A — 2 L of water A per day
  Arms: Water A
Dietary Supplement: Water B — 2 L of water B per day
  Arms: Water B

SUMMARY:
Evaluation of changes in skin metabolism after one month of intake of Acqua Rocchetta (water A) vs bicarbonate-calcic mediomineral water (water B) (reprogramming effect on skin metabolism); Evaluation of urinary profiles after intake of Acqua Rocchetta (water A) vs bicarbonate-calcic mediomineral water (water B) and possible relation with skin metabolites.

DETAILED DESCRIPTION:
This is a single-center, interventional, randomized controlled clinical trial conducted in healthy volunteers, in a double blind (subject and investigator).

The study will include age-matched female subjects who blindly take water A or water B, both marketed as food and not supplements, therefore evaluated annually by the relevant bodies (ASL, NAS and the Central Inspectorate for quality protection. and the repression of fraud on agri-food products (Icqrf)).

Women between 30 and 50 years old will be chosen who have a skin aging pattern very different from the male sex and governed by the oscillations of the menstrual cycle. A positive result on this population would be of crucial importance in terms of nutriceuticals and generalizability.

ELIGIBILITY:
Inclusion Criteria:

* healthy female subjects
* in good health without disease with an ICD code in compliance with the World Health Organisation definition (a state of complete physical, mental and social well-being and not merely the absence of disease or infirmity." )
* abstemious
* individuals who agree to sign an informed consent form
* individuals who follow an omnivorous diet

Exclusion Criteria:

* subjects outside the age range considered
* smokers and/or those with chronic or acute diseases coded by the ICD-10 system
* persons who do not consent to sign the informed consent form
* subjects who follow diets that are not omnivorous or with fattening / slimming purposes
* subjects undergoing hormonal or contraceptive hormonal therapies or in general drugs that may alter the hydroelectric balance
* persons with significant alterations in the menstrual cycle (amenorrhoea or dysmenorrhoea).
* use of alcohol.
* pregnancy (verified by self-declaration) and/or breastfeeding
* allergy to the components of Leukopor

Ages: 30 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Estimated)
Dates: Start 2021-06-29 (Actual); Primary Completion 2021-09 (Estimated); Study Completion 2021-09 (Estimated)

PRIMARY OUTCOMES:
Lipidomics | three months
  Different concentration in cutaneous lipids

SECONDARY OUTCOMES:
Urinomics | three months
  quantfication of different urinary metabolites

CONTACTS AND LOCATIONS:
Overall Officials: Paolo Pigatto, Prof, Principal Investigator — IRCSS Istituto Ortopedico Galeazzi
Locations (1):
- IRCSS Istituto Ortopedico Galeazzi, Milan, Italy

IPD SHARING:
Plan to Share IPD: No